CLINICAL TRIAL: NCT06230848
Title: Multisensory Early Oral Administration of Human Milk in Preterm Infants to Attenuate Early Life Toxic Stress on Epigenetic Modifications and Dysbiosis: Randomized Controlled Trial Pilot Study
Brief Title: Multisensory Early Oral Administration of Human Milk in Preterm Infants
Acronym: M-MILK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Thao Griffith, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 217411
Record Dates: First submitted 2024-01-05; First posted 2024-01-30 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Infant Development; Stress
Keywords: stress; preterm infants; epigenetics; gut microbiome; parent-infant relationship

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Infants in the control group will receive standard of care.
- M-MILK (Experimental): Infants in the M-MILK group will receive the M-MILK intervention in addition to standard of care.
  Interventions: Other: Multisensory Early Oral Administration of Human Milk (M-MILK)

INTERVENTIONS:
Other: Multisensory Early Oral Administration of Human Milk (M-MILK) — M-MILK is implemented starting on day 3 of life, after every hands-on care, during the beginning of a full gavage feeding. Infants receive M-MILK in small droplets via a 1-ml syringe. M-MILK will cease upon oral feeding initiation. Infants will receive either mother's own milk or donor's milk based on availability. Infants may receive up to 1 mL of milk each time based on their cues and responses. The 1 mL volume intake is included as part of their oral caloric intake. M-MILK is provided by nurses or parents.
  Arms: M-MILK

SUMMARY:
The aims of this pilot are to determine the feasibility and acceptability of the Multisensory early oral administration of human milk (M-MILK) intervention, recruitment, retention, and obtain data for sample size estimation. This study will advance nursing science and practice because it will inform our R01 RCT to examine the efficacy of M-MILK to attenuate adverse effects of early life toxic stress in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* born between 22 to 34 weeks gestational age and receiving mother's own milk and/or donor milk.

Exclusion Criteria:

* receiving only formula, oral cavity defects, gastrointestinal defects, chromosomal abnormalities, severe cardiac defects that require surgery, or intraventricular hemorrhage grade III or IV

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Chicago, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Attention Control: Infants in the attention control group will receive standard of care.
Period: Overall Study
Arm/Group | Attention Control | M-MILK
Started | 4 | 10
Completed | 4 | 7
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Population: Enrolled and completed baseline assessments
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Control | M-MILK | Total
Number analyzed (Participants) | 4 | 10 | 14
Age, Continuous [Median (Full Range); unit: weeks] — Gestational age at birth measured in weeks
  weeks | 30.5 [27 to 31] | 27 [23 to 30] | 27 [23 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Black | 0 | 4 | 4
  Non-Hispanic White | 2 | 3 | 5
  Hispanic | 1 | 3 | 4
  Non-Hispanic Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 10 | 14
Birthweight [Median (Full Range); unit: grams] — Birthweight in grams
  grams | 1525 [999 to 1865] | 875 [490 to 1585] | 977 [490 to 1865]
Small for gestational age [Count of Participants; unit: Participants] | 0 | 2 | 2
Intrauterine growth restriction [Count of Participants; unit: Participants] | 0 | 3 | 3
Preterm premature rupture of the membranes [Count of Participants; unit: Participants] — Population: Baseline measure was unavailable for one participant
  Participants
    number analyzed (Participants) | 4 | 9 | 13
    (all) | 1 | 7 | 8

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention
Description: The count of participants who receive M-MILK in at least 50% of their scheduled M-MILK administrations. MILK will be considered feasible if M-MILK is implemented by nurses or parents after every hands-on care and during the beginning of a full gavage feeding at least 50% of the time.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Population: Only the intervention arm is assessed for feasibility.
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 0 | 10
Participants | 0 | 7

2. Primary Outcome: Acceptability of Intervention
Description: The percentage of parents who rate the intervention as very positive, slightly positive, or acceptable on a 5-point Likert scale.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Population: Reported by the parent in the study exit survey. Only parents in the M-MILK group were asked about the intervention. Two parents did not complete the acceptability survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 0 | 5
Participants | 0 | 5

3. Primary Outcome: Retention
Description: Retention will be described by the number of post-discharge follow-up surveys completed.
Time Frame: 2 months corrected age
Measure: Count of Participants; unit: Participants
Groups:
- M-MILK: Infants in the M-MILK group will receive the M-MILK intervention in addition to standard of care.
  Multisensory Early Oral Administration of Human Milk (M-MILK): M-MILK is implemented starting on day 3 of life, during the day shift, after every hands-on care, during the beginning of a full gavage feeding. Infants receive M-MILK in small droplets via a 1-ml syringe. M-MILK will cease upon oral feeding initiation. Infants will receive either mother's own milk or donor's milk based on availability. Infants may receive up to 1 mL of milk each time based on their cues and responses. The 1 mL volume intake is included as part of their oral caloric intake. M-MILK is provided by nurses or parents.
Arm/Group | Control | M-MILK
Number analyzed (Participants) | 4 | 10
Participants | 4 | 7

4. Primary Outcome: The Scarf Sign Cluster of the Neurobehavioral Assessment of the Preterm Infants Score
Description: The Neurobehavioral Assessment of the Preterm Infants (NAPI, 73 items, 32-37 weeks PMA): cluster score for scarf sign ranges from 0-100, where higher scores indicate better neurodevelopmental performance.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 4 | 7
score on a scale | 66.7 [66.7 to 66.7] | 66.7 [66.7 to 66.7]

5. Primary Outcome: Variability in the Motor Development & Vigor Cluster of the Neurobehavioral Assessment of the Preterm Infants Score
Description: The Neurobehavioral Assessment of the Preterm Infants (NAPI, 73 items, 32-37 weeks PMA): cluster score for motor development & vigor ranges from 0-100, where higher scores indicate better neurodevelopmental performance.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 4 | 7
score on a scale | 53.1 [41.3 to 70.4] | 60.9 [49.2 to 75.0]

6. Primary Outcome: Popliteal Angle Cluster of the Neurobehavioral Assessment of the Preterm Infants Score
Description: The Neurobehavioral Assessment of the Preterm Infants (NAPI, 73 items, 32-37 weeks PMA): cluster score for popliteal angle ranges from 0-100, where higher scores indicate better neurodevelopmental performance.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 4 | 7
score on a scale | 16.7 [0 to 66.7] | 66.7 [0 to 100]

7. Primary Outcome: Alertness and Orientation Cluster of the Neurobehavioral Assessment of the Preterm Infants Score
Description: The Neurobehavioral Assessment of the Preterm Infants (NAPI, 73 items, 32-37 weeks PMA): cluster score for alertness and orientation ranges from 0-100, where higher scores indicate better neurodevelopmental performance.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 4 | 7
score on a scale | 41.3 [7.5 to 69.1] | 82.5 [25.4 to 85.7]

8. Primary Outcome: Irritability Cluster of the Neurobehavioral Assessment of the Preterm Infants Score
Description: The Neurobehavioral Assessment of the Preterm Infants (NAPI, 73 items, 32-37 weeks PMA): cluster score for irritability ranges from 0-100, where higher scores indicate better neurodevelopmental performance.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 4 | 7
score on a scale | 33.4 [16.7 to 33.4] | 33.4 [0 to 36.9]

9. Primary Outcome: Quality of Cry Cluster of the Neurobehavioral Assessment of the Preterm Infants Score
Description: The Neurobehavioral Assessment of the Preterm Infants (NAPI, 73 items, 32-37 weeks PMA): cluster score for quality of cry ranges from 0-100, where higher scores indicate better neurodevelopmental performance.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Population: Cry quality is only measured if the infant was crying during the assessment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 3 | 4
score on a scale | 0 [0 to 33.3] | 25 [0 to 75]

10. Primary Outcome: Percent Sleep Cluster of the Neurobehavioral Assessment of the Preterm Infants Score
Description: The Neurobehavioral Assessment of the Preterm Infants (NAPI, 73 items, 32-37 weeks PMA): cluster score for percent sleep ranges from 0-100, where higher scores indicate better neurodevelopmental performance.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 4 | 7
score on a scale | 14.3 [7.1 to 57.1] | 14.3 [0 to 57.1]

11. Primary Outcome: Early Feeding Skill Assessment Score
Description: EFS has 22 items (32-50 weeks PMA), summary scores, 5 subscales: respiratory regulation (range 5 - 15), oral-motor functioning (range 4 - 12), swallowing coordination (range 4 - 12), engagement (range 2 - 6), & physiologic stability (range 4 - 12), where higher scores indicate better oral feeding skill development. The total score is the sum of the subscales and ranges from 19-57.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- M-MILK: Infants in the M-MILK group will receive the M-MILK intervention in addition to standard of care.
  Multisensory Early Oral Administration of Human Milk (M-MILK): M-MILK is implemented starting on day 3 of life, during the day shift, after every hands-on care, during the beginning of a full gavage feeding, and up to 4 times a day. Infants receive M-MILK in small droplets via a 1-ml syringe. M-MILK will cease upon oral feeding initiation. Infants will receive either mother's own milk or donor's milk based on availability. Infants may receive up to 1 mL of milk each time based on their cues and responses. The 1 mL volume intake is included as part of their oral caloric intake. M-MILK is provided by nurses or parents.
Arm/Group | Control | M-MILK
Number analyzed (Participants) | 4 | 7
score on a scale | 47.3 (3.9) | 49.6 (5.3)

12. Secondary Outcome: Parent Stressor Scale: NICU Score
Description: Scores range from 1 to 5, where higher scores indicate greater parental stress..
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Population: Two parents in the M-MILK group did not complete this survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- M-MILK: Infants in the M-MILK group will receive the M-MILK intervention in addition to standard of care.
  Multisensory Early Oral Administration of Human Milk (M-MILK): M-MILK is implemented as droplets, at day 3 of life, after every hands-on care, and during the beginning of a full gavage feeding. The infant may be supportively positioned in bed, held skin-to-skin by caregiver, or held/cradled by nurse or caregiver. The nurse draws up 1 mL of milk into the 1-mL syringe from a prepared bottle or enteral feeding syringe. The nurse then proceeds to implement M-MILK while observing the infant's responses closely. The nurse talks to the infant with a soft calm voice while providing gentle touch throughout the intervention. The nurse begins M-MILK by first placing 1-2 drops of milk onto the infant's upper lip, allowing the infant to feel and smell the milk. The nurse gently strokes the infant's lips with a pacifier/swab or infant's fingers. M-MILK will be provided based on infants' responses and cues. M-MILK is concluded if the infant is no longer engaged or has finished the 1 mL of milk.
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 4 | 5
score on a scale | 2.4 (1.2) | 2.3 (1.0)

13. Secondary Outcome: Parent Discharge Readiness Score
Description: Scores range from 44 to 308, where higher scores indicate more parental readiness for discharge.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 4 | 6
score on a scale | 231.0 [199.5 to 246.5] | 211.0 [206.0 to 246.0]

14. Secondary Outcome: Breastmilk Pumping Rate
Description: The percentage of mothers who report breastmilk pumping at discharge.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Population: Two parents in the M-MILK group did not report this data at discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 4 | 5
Participants | 1 | 5

15. Secondary Outcome: Breastfeeding Rate
Description: The percentage of mothers who report breastfeeding at discharge.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 3 | 3
Participants | 0 | 1

16. Secondary Outcome: Maternal Edinburgh Postnatal Depression Scale Score
Description: Scores range from 0 to 30, where higher scores indicate greater depressive symptoms
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Population: Two parents in the M-MILK group did not complete this survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attention Control | M-MILK
Number analyzed (Participants) | 4 | 5
score on a scale | 3.8 (4.5) | 4.8 (4.9)

17. Other Pre Specified Outcome: Variability in Gut Microbial Community Structure and Relative Abundance of SCFA- and Lactate- Producing Bacteria
Description: Alpha diversity indices will be obtained. Differential abundance individual taxa will be obtained.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Variability in DNA Methylation of NR3C1 Promoter
Description: The percent DNAm at the NR3C1 promoters and at each CpG site will be quantified.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Variability in DNA Methylation of HSD11B2 Promoter
Description: The percent DNAm at the HSD11B2 promoters and at each CpG site will be quantified.
Time Frame: At the time of discharge from NICU, which is typically 10 to 16 weeks from birth.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated from randomization to hospital discharge, which is typically 10 to 16 weeks from birth.
Arm/Group | Attention Control | M-MILK
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/10
Other Adverse Events (participants affected / at risk) | 0/4 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT06230848/Prot_SAP_000.pdf